CLINICAL TRIAL: NCT07374536
Title: Clinical and Radiographic Evaluation of Local Application of Melatonin on Postoperative Outcomes After Surgical Removal of Impacted Mandibular Third Molar: A Randomized Controlled Study
Brief Title: Clinical and Radiographic Evaluation of Local Application of Melatonin on Postoperative Outcomes After Surgical Removal of Impacted Mandibular Third Molar
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/1006
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Impact Molar
Keywords: Impaction; Melatonin; Mandibular 3rd Molars; Radiographic evaluation; Clinical Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control without Melatonin (Placebo Comparator): (the extraction socket will be left empty followed by suture of the socket after extraction
  Interventions: Diagnostic Test: Control; Dietary Supplement: Melatonin gel
- Study with Melatonin (Experimental): 3 mg of melatonin into 2 ml of 2% hydroxyethyl cellulose gel will be packed into the socket after extraction
  Interventions: Diagnostic Test: Control; Dietary Supplement: Melatonin gel

INTERVENTIONS:
Diagnostic Test: Control — the extraction socket will be left empty followed by suture of the socket after extraction
Dietary Supplement: Melatonin gel — 3 mg of melatonin into 2 ml of 2% hydroxyethyl cellulose gel will be packed into the socket after extraction

SUMMARY:
Clinical and Radiographic Evaluation of Local Application of Melatonin on Postoperative Outcomes after Surgical Removal of Impacted Mandibular Third Molar: A Randomized Controlled Study

DETAILED DESCRIPTION:
of all impacted teeth. The frequency of impaction of the mandibular third molar ranges from 33% to 58.7% (Breik O and Grubor D.,2008). A tooth is considered to be impacted when its eruption time has passed or when the eruption interferes with the normal functional occlusion with other teeth or the overlying bone or soft tissues in the oral cavity (Celikoglu et al.,2010)).

The surgical removal of an impacted third molar is an everyday procedure in oral surgery clinics. However, it is known to disturb the quality of life of the patient by restricting the ability to chew food, open the mouth, and speak (Lago-Mendez et al., 2007). Furthermore, there is a danger of periodontal damage on the distal root of the adjacent molar which could affect healing (Richardson et al., 2005), 43% of the patients had a periodontal pocket depth of 7 mm or more at the distal root of the mandibular second molar 2 years post extraction of an impacted mandibular third molar.

The healing of periodontal defects related to the distal root of the adjacent molar may be compromised by intra-bony defects and bone loss after the removal of the impacted tooth. Alternative strategies, such as different flap designs, soft-tissue suturing, socket preservation, and tissue regeneration techniques with autologous bone, allografts, xenografts, or alloplastic grafts, have been proposed to prevent periodontal defects and physiological bone resorption after the surgical extraction of the mandibular third molar (Toledano-Serrabona et al.,2021).

Melatonin is a growth hormone secreted mainly by the pineal gland and other structures, such as the retina, skin, gastrointestinal tract, lymphocytes, and bone marrow (Radogna et al.,2010).It has antioxidant and anti inflammatory properties. It inhibits the production of reactive oxidants by reducing the expression of cyclooxygenase-2 and prostaglandin. In addition, it attracts polymorphonuclear cells to the site of injury (Cutando et al.,2007).

ELIGIBILITY:
Inclusion Criteria: 1)Both genders are included. 2)Adult patients (18-40) years 3)Healthy American Society of Anesthesiologists ASA I Patients. 4)Patients with class I or II impacted lower third molars with position A or B.

-

Exclusion Criteria:

1. Pregnant & lactating women.
2. Smoker patients.
3. Patients with poor oral hygiene.
4. Patients with bad oral habits as bruxism.
5. Patients with periapical or peri coronal lesions.
6. Patients with aggressive gingivitis or periodontitis.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Bone density | 1 and 4 months postoperatively
  Assess relative bone density at the center of the extracted socket using digital periapical radiograph in the center of the socket.

SECONDARY OUTCOMES:
Post-operative pain levels | 1, 3 and 7 days Postoperatively
  Post-operative pain levels by VAS (Visual Analog Scale)
Measure Edema scale | 1, 3 and 7 days Postoperatively
  Measure Edema scale using flexible ruler
Measure Maximal Mouth opening (MMO) | 1, 3 and 7 days Postoperatively
  Measure Maximal Mouth opening (MMO) using digital caliper.
Measure the incidence of post-operative complications | 1, 3 and 7 days Postoperatively
  Measure the incidence of post-operative complications (e.g., dry socket, infection) in both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Suez Canal University, Ismailia, Egypt, Egypt